CLINICAL TRIAL: NCT02348034
Title: A Randomized Controlled Trial Exploring the Ability of Negative Pressure Wound Therapy (NPWT) to Reduce Colorectal Surgical Site Infections (SSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Kinetic Concepts, Inc. (Industry); Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Gary Groot, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-259
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Site Infection (SSI); Negative Pressure Wound Therapy (NPWT)
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevena Dressing (Experimental): This group will receive prevena dressing after the elective colorectal surgery
  Interventions: Device: Prevena Dressing
- Conventional dressing (No Intervention): This group will receive conventional dressing after the elective colorectal surgery

INTERVENTIONS:
Device: Prevena Dressing — Prevena dressing will be applied to the closed surgical wound after the elective colorectal surgery to evaluate its ability to reduce surgical site infections.
  Arms: Prevena Dressing

SUMMARY:
The study will explore the ability of negative pressure wound therapy (Prevena dressing) to reduce post operative superficial surgical site infection rate in elective colorectal surgery. Half of the participants will receive Prevena dressing on closed incision immediately after the operation while other half will receive conventional surgical dressing.

DETAILED DESCRIPTION:
The trial will commence with recruitment of participants after an assessment of their potential eligibility. Those recruited in the trial will sign informed consent either on the day of surgery or during the PAC appointment, before any study-related activities are performed.

Perioperative measures will include bowel preparation with Fleet Phospho-soda, preoperative shaving with electric clippers 1 hour before the operation, and intravenous prophylactic antibiotic administered 30 minutes before the incision, and repeated in OR if the operation lasts more than 3 hours, and discontinued within 24 h after the operation. In all procedures, chlorhexidine solution will be applied to the skin to achieve preoperative skin antisepsis, and the usual reusable or disposable surgical gowns, drapes, and gloving will be used. The type of surgical procedure will be a colorectal resection for any malignant or benign condition of the colon, rectum or anal canal via a laparotomy wound. The type of incision will either be a vertical midline or transverse abdominal incision. Laparotomy wound will be closed primarily as a mass closure technique utilizing polydioxanone (PDS) or Nylon suture. Skin and subcutaneous tissues will be approximated using stainless-steel staples.

During the surgery, assessment of eligibility (including wound classification) will be completed, and if eligible, the participant will be randomized to one of the two treatment arms - group A (conventional dressing) or group B (Prevena dressing). The randomization scheme is described later in the protocol. After the surgical wound is closed, the assigned dressing - conventional dressing (Mepore) or Prevena dressing - will be applied.

For participants in group A (conventional dressing) the wound will be inspected on an as needed basis during postoperative days 1-6 to assess for SSI (where day 0 = day of surgery). On postoperative day 7, the dressing will be removed. If the participant is in hospital, the wound care nurse or study staff will remove the dressing and examine the wound for SSI. If the participant was discharged before postoperative day 7, the home care nurse or the participant's physician will remove the dressing. The patient will have been sent home with a Post-Op Day 7 follow-up form, and will have been instructed to provide the form to the home care nurse or their physician to complete for the assessment for SSI.

For participants randomized to group B (Prevena dressing), the wound care nurse or study staff will inspect the dressing daily during postoperative days 1-6 (where day 0 = day of surgery) to assess for proper functioning of the Prevena dressing. If the participant is discharged before postoperative day 7, the wound care nurse or study staff will contact the participant daily to check for proper functioning of the Prevena dressing. On postoperative day 7, the Prevena dressing will be removed. If the participant is in hospital, the wound care nurse or study staff (residents or Surgeons) will remove the dressing and assess the wound for SSI. If the participant was discharged before postoperative day 7, the home care nurse or the participant's physician will remove the dressing. The patient will have been sent home with a Post-Op Day 7 follow-up form, and will have been instructed to provide the form to the home care nurse or their physician to complete for signs of SSI.

If SSI is suspected, the participant will be advised to visit the clinic for assessment of SSI by the study team. In case it is not possible for the participant to visit the clinic for assessment of SSI by the study team, the participants will have been sent home with a SSI Confirmation form to be completed by the participant's physician.

The wound care nurse or study staff will conduct post-discharge follow-up on postoperative days 14 (± 2 days) and 21 (± 2 days) by telephoning the family physician or the participant to check whether there are signs of SSI. If SSI is suspected, the participant will be advised to visit the clinic for assessment of SSI by the study team. If not possible, the participant will be instructed to ask their physician to complete the SSI Confirmation form.

On postoperative day 30 (± 7 days), the participant will be seen in the clinic by the treating surgeon as a part of the treatment and follow-up plan, and the wound will be assessed for SSI. For participants who are not able to come to the clinic, the study team will contact the participant or the family physician by telephone to check whether there are signs of SSI. If SSI is suspected, the participant will be advised to visit the clinic for assessment of SSI by the study team. If not possible, the participant will be instructed to ask their physician to complete the SSI Confirmation form.

As described above, each participant will have up to 12 study visits (11 scheduled visits, including the day of surgery, plus one clinic visit if there is suspicion of SSI). At any point, however, once SSI is confirmed, the participant will undergo no further study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 18 years
2. Patient undergoing colorectal resective surgery for any reason (benign or malignant) such as diverticular disease, colorectal cancer or inflammatory bowel disease through a laparotomy wound
3. Class II surgical wound
4. Laparoscopically assisted colorectal procedure

Exclusion Criteria:

1. Patient requires emergent or urgent operation
2. Patient has advanced colorectal malignancy associated with peritoneal carcinomatosis
3. Class III or IV surgical wound
4. Laparoscopic surgery involving intracorporeal colorectal resection and anastomosis
5. Patient has a previous disfigured midline laparotomy surgical scar requiring wide excision of skin, subcutaneous tissue, fascia and muscle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Presence/Absence of superficial surgical site infection | Postoperative day 30.
  Primary outcome of interest will be the presence and/or absence of superficial surgical site infection at postoperative day 30.

SECONDARY OUTCOMES:
Presence/Absence of intervention related side effects | Postoperative day 30.
  The secondary outcome will be any side effects related to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Groot, Principal Investigator — University of Saskatchewan
Locations (3):
- Canada (3):
  - St. Paul's Hospital, 1081 Burrard Street, C310, Vancouver, British Columbia
  - St. Paul's Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Measures displayed on Hospital Compare. 2013. Available at: http://www.medicare.gov/hospitalcompare/ Data/Measures-Displayed.html. Accessed March 22, 2013
- [Background] Wick EC, Vogel JD, Church JM, Remzi F, Fazio VW. Surgical site infections in a "high outlier" institution: are colorectal surgeons to blame? Dis Colon Rectum. 2009 Mar;52(3):374-9. doi: 10.1007/DCR.0b013e31819a5e45. PMID 19333034
- [Background] Anthony T, Murray BW, Sum-Ping JT, Lenkovsky F, Vornik VD, Parker BJ, McFarlin JE, Hartless K, Huerta S. Evaluating an evidence-based bundle for preventing surgical site infection: a randomized trial. Arch Surg. 2011 Mar;146(3):263-9. doi: 10.1001/archsurg.2010.249. Epub 2010 Nov 15. PMID 21079110
- [Background] Tang R, Chen HH, Wang YL, Changchien CR, Chen JS, Hsu KC, Chiang JM, Wang JY. Risk factors for surgical site infection after elective resection of the colon and rectum: a single-center prospective study of 2,809 consecutive patients. Ann Surg. 2001 Aug;234(2):181-9. doi: 10.1097/00000658-200108000-00007. PMID 11505063
- [Background] Smith RL, Bohl JK, McElearney ST, Friel CM, Barclay MM, Sawyer RG, Foley EF. Wound infection after elective colorectal resection. Ann Surg. 2004 May;239(5):599-605; discussion 605-7. doi: 10.1097/01.sla.0000124292.21605.99. PMID 15082963
- [Background] Smyth ET, Emmerson AM. Surgical site infection surveillance. J Hosp Infect. 2000 Jul;45(3):173-84. doi: 10.1053/jhin.2000.0736. PMID 10896795
- [Background] Weiss CA 3rd, Statz CL, Dahms RA, Remucal MJ, Dunn DL, Beilman GJ. Six years of surgical wound infection surveillance at a tertiary care center: review of the microbiologic and epidemiological aspects of 20,007 wounds. Arch Surg. 1999 Oct;134(10):1041-8. doi: 10.1001/archsurg.134.10.1041. PMID 10522843
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Martone WJ, Nichols RL. Recognition, prevention, surveillance, and management of surgical site infections: introduction to the problem and symposium overview. Clin Infect Dis. 2001 Sep 1;33 Suppl 2:S67-8. doi: 10.1086/321859. No abstract available. PMID 11486301
- [Background] Gaynes RP, Culver DH, Horan TC, Edwards JR, Richards C, Tolson JS. Surgical site infection (SSI) rates in the United States, 1992-1998: the National Nosocomial Infections Surveillance System basic SSI risk index. Clin Infect Dis. 2001 Sep 1;33 Suppl 2:S69-77. doi: 10.1086/321860. PMID 11486302
- [Background] Astagneau P, Rioux C, Golliot F, Brucker G; INCISO Network Study Group. Morbidity and mortality associated with surgical site infections: results from the 1997-1999 INCISO surveillance. J Hosp Infect. 2001 Aug;48(4):267-74. doi: 10.1053/jhin.2001.1003. PMID 11461127
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Background] Measures displayed on Hospital Compare. 2013. Available at: ttp://www.medicare.gov/hospitalcompare /Data/Measures-Displayed.html. Accessed March 22, 2013.
- [Background] Stulberg JJ, Delaney CP, Neuhauser DV, Aron DC, Fu P, Koroukian SM. Adherence to surgical care improvement project measures and the association with postoperative infections. JAMA. 2010 Jun 23;303(24):2479-85. doi: 10.1001/jama.2010.841. PMID 20571014
- [Background] Fujii T, Tabe Y, Yajima R, Yamaguchi S, Tsutsumi S, Asao T, Kuwano H. Effects of subcutaneous drain for the prevention of incisional SSI in high-risk patients undergoing colorectal surgery. Int J Colorectal Dis. 2011 Sep;26(9):1151-5. doi: 10.1007/s00384-011-1228-2. Epub 2011 May 7. PMID 21553008
- [Background] Reid K, Pockney P, Draganic B, Smith SR. Barrier wound protection decreases surgical site infection in open elective colorectal surgery: a randomized clinical trial. Dis Colon Rectum. 2010 Oct;53(10):1374-80. doi: 10.1007/DCR.0b013e3181ed3f7e. PMID 20847618
- [Background] Edwards JP, Ho AL, Tee MC, Dixon E, Ball CG. Wound protectors reduce surgical site infection: a meta-analysis of randomized controlled trials. Ann Surg. 2012 Jul;256(1):53-9. doi: 10.1097/SLA.0b013e3182570372. PMID 22584694
- [Background] Aimaq R, Akopian G, Kaufman HS. Surgical site infection rates in laparoscopic versus open colorectal surgery. Am Surg. 2011 Oct;77(10):1290-4. doi: 10.1177/000313481107701003. PMID 22127072
- [Background] Schwenk W, Haase O, Neudecker J, Muller JM. Short term benefits for laparoscopic colorectal resection. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003145. doi: 10.1002/14651858.CD003145.pub2. PMID 16034888
- [Background] Kang CY, Halabi WJ, Luo R, Pigazzi A, Nguyen NT, Stamos MJ. Laparoscopic colorectal surgery: a better look into the latest trends. Arch Surg. 2012 Aug;147(8):724-31. doi: 10.1001/archsurg.2012.358. PMID 22508667
- [Background] Gomoll AH, Lin A, Harris MB. Incisional vacuum-assisted closure therapy. J Orthop Trauma. 2006 Nov-Dec;20(10):705-9. doi: 10.1097/01.bot.0000211159.98239.d2. PMID 17106382
- [Background] Reddix RN Jr, Leng XI, Woodall J, Jackson B, Dedmond B, Webb LX. The effect of incisional negative pressure therapy on wound complications after acetabular fracture surgery. J Surg Orthop Adv. 2010 Summer;19(2):91-7. PMID 20727304
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Fleischmann W, Lang E, Russ M. [Treatment of infection by vacuum sealing]. Unfallchirurg. 1997 Apr;100(4):301-4. doi: 10.1007/s001130050123. German. PMID 9229781
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Suissa D, Danino A, Nikolis A. Negative-pressure therapy versus standard wound care: a meta-analysis of randomized trials. Plast Reconstr Surg. 2011 Nov;128(5):498e-503e. doi: 10.1097/PRS.0b013e31822b675c. PMID 22030509
- [Background] Colli A, Camara ML. First experience with a new negative pressure incision management system on surgical incisions after cardiac surgery in high risk patients. J Cardiothorac Surg. 2011 Dec 6;6:160. doi: 10.1186/1749-8090-6-160. PMID 22145641
- [Background] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Background] Benech A, Arcuri F, Poglio G, Brucoli M, Guglielmetti R, Crespi MC, Pia F. Vacuum-assisted closure therapy in reconstructive surgery. Acta Otorhinolaryngol Ital. 2012 Jun;32(3):192-7. PMID 22767986
- [Background] Orgill DP, Manders EK, Sumpio BE, Lee RC, Attinger CE, Gurtner GC, Ehrlich HP. The mechanisms of action of vacuum assisted closure: more to learn. Surgery. 2009 Jul;146(1):40-51. doi: 10.1016/j.surg.2009.02.002. Epub 2009 Apr 19. No abstract available. PMID 19541009
- [Background] Guidance for Industry. Chronic Cutaneous Ulcer and Burn Wounds-Developing Products for Treatment (Draft Guidance). Rockville,MD, U.S. Department of Health and Human Services, 2000, p. 15
- [Background] Surgical Site Infection (SSI) Event. Centers for Disease Control, 2015